CLINICAL TRIAL: NCT04773392
Title: SIMPLE Study: A Prospective and Randomized Trial of a Simplified Immunosuppressive Protocol Utilizing Low Dose EnvarsusXR
Brief Title: Simplified IMmunosuppressive Protocol Utilizing Low Dose EnvarsusXR
Acronym: SIMPLE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Research contract expired
Sponsor: University of Southern California (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Santhi Voora, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-18-00513
Record Dates: First submitted 2021-02-15; First posted 2021-02-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation; Kidney Transplant Rejection
Keywords: tacrolimus; envarsus XR; kidney transplant; rejection; immunosuppressive agents; renal transplant
MeSH Terms: conditions — Rejection, Psychology | interventions — Basiliximab; Methylprednisolone; Prednisone; Steroids; Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, prospective clinical trial. Patients will be screened prior to surgery and randomized 1:1 to each arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Twice-daily Regimen (Active Comparator): Twice-daily regimen of immediate release tacrolimus, mycophenolate mofetil (MMF)/mycophenolic acid (MPA) plus daily methylprednisolone or prednisone.
  Interventions: Drug: Twice-daily Tacrolimus; Drug: Induction Immunosuppression with Basiliximab or Rabbit Anti Thymoglobulin (rATG); Drug: Methylprednisolone, prednisone; Drug: Mycophenolate mofetil (MMF) or Mycophenolic acid (MPA)
- Once-daily Regimen (Active Comparator): Once-daily regimen of Envarsus, azathioprine plus methylprednisolone or prednisone.
  Interventions: Drug: Once-daily envarsus XR; Drug: Induction Immunosuppression with Basiliximab or Rabbit Anti Thymoglobulin (rATG); Drug: Methylprednisolone, prednisone; Drug: Azathioprine

INTERVENTIONS:
Drug: Twice-daily Tacrolimus — Within 48 hours of transplantation, immediate release tacrolimus (IRT) (0.1 mg/kg /day) will be administered twice a day.
  Other Names: immediate release tacrolimus
  Arms: Twice-daily Regimen
Drug: Once-daily envarsus XR — Within 48 hours of transplantation, Envarsus XR (0.13mg/kg/day) will be administered once a day.
  Other Names: extended releated tacrolimus
  Arms: Once-daily Regimen
Drug: Induction Immunosuppression with Basiliximab or Rabbit Anti Thymoglobulin (rATG) — Induction immunosuppression with Basiliximab or Rabbit Anti Thymoglobulin (rATG) per protocol. The dose of Basiliximab will be a standard of two 20 mg doses and total rATG will not exceed 6 mg/kg.
  Other Names: Simulect, ATG
Drug: Methylprednisolone, prednisone — Methylprednisolone intraoperatively (500mg) and immediately post transplantation (200mg on post operative day (POD) #1, 150mg on POD#2, 100mg on POD#3) then oral prednisone (50mg on POD #4, 20mg on POD #5). Oral prednisone will be tapered down to a minimal dose of 5mg within 6 weeks post transplantation.
  Other Names: Steroids
Drug: Mycophenolate mofetil (MMF) or Mycophenolic acid (MPA) — Mycophenolate mofetil (MMF) (up to 1000mg) or Mycophenolic acid (MPA) (up to 720mg) will be administered twice a day.
  Other Names: Twice a day anti-metabolite
  Arms: Twice-daily Regimen
Drug: Azathioprine — Azathioprine (1-3 mg/kg) will be administered once a day.
  Other Names: Once a day anti-metabolite
  Arms: Once-daily Regimen

SUMMARY:
The purpose of this study is to determine if the combination of once-daily tacrolimus extended-release (EnvarsusXR) and Azathioprine is non inferior with respect to the composite outcome of acute rejection, graft and patient survival as compared to a combination of twice-daily immediate release tacrolimus and mycophenolate mofetil/mycophenolic acid.

DETAILED DESCRIPTION:
While short-term graft outcomes in kidney transplantation have improved, this requires adherence to a complex medication regimen. The current twice-daily immunosuppressive regimen, immediate release tacrolimus and mycophenolate mofetil/mycophenolic acid, has reduced rejection rates significantly, but frequently cause neurologic and gastrointestinal side effects which impact recipient quality of life. These side effects often require dose adjustments and studies have shown inferior outcomes when multiple changes are made to the immunosuppressive regimen. Furthermore, patients taking twice-daily medications have poorer compliance and yet adherence to these medications is critical to mitigate the risk of allograft rejection. Acute and chronic rejection are important causes of graft failure and patient survival.

Immediate release (IR) tacrolimus based immunosuppressive regimens have become the standard of care at most US centers. With the introduction of a once-daily tacrolimus formulation, kidney transplant recipients can now be on a combination regimen (EnvarsusXR and azathioprine) that permits all immunosuppressive medications to be taken once a day instead of twice . Previous studies suggest that therapeutic goals with EnvarsusXR may be achieved at a lower dose than the currently recommended dose. This once a day medication schedule has the potential to simplify the immunosuppressive regimen by reducing adverse side effects and facilitating compliance.

The investigators seek to demonstrate that a once-daily regimen, including EnvarsusXR and azathioprine, will be at least equally effective with respect to acute rejection, graft and patient survival as compared to the standard, twice-daily, immediate release tacrolimus and mycophenolate mofetil/mycophenolic acid. The investigators will also assess graft function, medication complications and side effects in each arm.

ELIGIBILITY:
Inclusion Criteria:

* De- Novo Kidney transplant patients between 18 and 85 years old
* Cold ischemia time (CIT) < 24 hours for 3-6 HLA mismatches between donor and recipient and CIT >24 hours for HLA mismatch of less than 3 between donor and recipient
* Most recent pre-transplant cPRA (calculated panel reactive antibody) ≤ 20%

Exclusion Criteria:

* Repeat kidney transplant recipients
* cPRA >20%
* rATG (rabbit anti-thymocyte globulin) induction >6mg/kg at time of induction
* Crossmatches deemed positive by accepting physician
* Presence of pre-formed anti-HLA (anti-Human Leukocyte Antigen) DSA (Donor-Specific Antibody) as defined by MFI (mean fluorescence intensity) approaching 3000 using flow cytometry/Luminex-based, specific anti-HLA antibody testing.
* Receipt of desensitization protocols
* History of skin cancer
* Recipient of multi-organ or dual kidney transplants
* For any condition, in which the investigator's opinion makes the subject unsuitable for study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
To compare the composite incidence of biopsy proven acute rejection, graft survival and patient survival | 3 months
  Biopsies will be performed for unexplained rise in serum creatinine or proteinuria and the development of donor specific antibodies. Biopsies will be assessed by a pathologist using standard Banff classification of renal allograft pathology. Graft loss will be defined as return to chronic dialysis or graft removal.
To compare the composite incidence of biopsy proven acute rejection, graft survival and patient survival | 6 months
  Biopsies will be performed for unexplained rise in serum creatinine or proteinuria and the development of donor specific antibodies. Biopsies will be assessed by a pathologist using standard Banff classification of renal allograft pathology. Graft loss will be defined as return to chronic dialysis or graft removal.
To compare the composite incidence of biopsy proven acute rejection, graft survival and patient survival | 12 months
  Biopsies will be performed for unexplained rise in serum creatinine or proteinuria and the development of donor specific antibodies. Biopsies will be assessed by a pathologist using standard Banff classification of renal allograft pathology. Graft loss will be defined as return to chronic dialysis or graft removal.

SECONDARY OUTCOMES:
Renal allograft function | Every month, for a duration of 12 months
  Estimated glomerular filtration rate (eGFR)
Proteinuria | Every month, for a duration of 12 months
  Urinalysis
Donor-specific antibodies (DSA) | 3, 6, and 12 months
  Donor-specific anti-HLA antibodies, with a MFI (mean fluorescence intensity) >1000, measured by flow cytometry/Luminex-based assay
Cytomegalovirus (CMV) | 3, 6, and 12 months
  CMV PCR
Liver Function | 3, 6, and 12 months
  Alanine aminotransferase, aspartate aminotransferase and alkaline phosphatase
Gastrointestinal side effects | 3, 6, and 12 months
  GI side effects will be assessed by the Gastrointestinal Symptoms Rating Scale (GSRS) is a 15 item questionnaire addressing reflux, abdominal pain, indigestion, diarrhea and constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Dyspepsia and quality of life | 3, 6, and 12 months
  The Quality of Life in Reflux and Dyspepsia (QOLRAD) is a 25 item instrument depicting problems with emotions, vitality, sleep, eating/drinking, and physical/social functioning in adult patients with reflux disease. The questions are rated on a seven-point graded Likert scale; lower values indicate a more severe impact on daily functioning.
Tremor | 3, 6, and 12 months
  Tremor will be assessed by Quality of life in Essential Tremor Questionnaire, (QUEST) a 30-item scale developed specifically for patients with essential tremor to measure items impacting perceived quality of life (QOL). The items are rated on a five-point scale (score 0-4), corresponding to the frequency (never, rarely, sometimes, frequently, always) with which tremor was perceived to currently impact a function or to be associated with various feelings and attitudes
Perception of quality of life | 3, 6, and 12 months
  The Short Form (36) Healthy Survey (SF-36) is a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being.Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Cancer | 3, 6, and 12 months
  Incidence of cancers
Diabetes | 3, 6, and 12 months
  Incidence of new onset diabetes measured by HgbA1c
Electrolytes | 3, 6, and 12 months
  Dose of magnesium, potassium and phosphorus needed to replete electrolytes
Adverse Events | 3, 6, and 12 months
  An adverse event can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use the product, whether or not related to the product.
Dose changes | 3, 6, and 12 months
  Frequency of dose changes made in Envarsus, tacrolimus and MMF/MPA. Dosage changes will be adjusted for Tacrolimus drug levels as per protocol. MMF/MPA will be adjusted depending on gastrointestinal tolerability and bone marrow suppression.
BK Viremia | 3, 6, 12 months
  BK quantitative serum assay

CONTACTS AND LOCATIONS:
Overall Officials: Santhi Voora, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park SI, Felipe CR, Pinheiro-Machado PG, Garcia R, Fernandes FB, Casarini DE, Tedesco-Silva H Jr, Medina-Pestana JO. Tacrolimus pharmacokinetic drug interactions: effect of prednisone, mycophenolic acid or sirolimus. Fundam Clin Pharmacol. 2009 Feb;23(1):137-45. doi: 10.1111/j.1472-8206.2008.00644.x. PMID 19267777
- [Background] Dalal P, Shah G, Chhabra D, Gallon L. Role of tacrolimus combination therapy with mycophenolate mofetil in the prevention of organ rejection in kidney transplant patients. Int J Nephrol Renovasc Dis. 2010;3:107-15. doi: 10.2147/ijnrd.s7044. Epub 2010 Aug 4. PMID 21694936
- [Background] Kulich KR, Madisch A, Pacini F, Pique JM, Regula J, Van Rensburg CJ, Ujszaszy L, Carlsson J, Halling K, Wiklund IK. Reliability and validity of the Gastrointestinal Symptom Rating Scale (GSRS) and Quality of Life in Reflux and Dyspepsia (QOLRAD) questionnaire in dyspepsia: a six-country study. Health Qual Life Outcomes. 2008 Jan 31;6:12. doi: 10.1186/1477-7525-6-12. PMID 18237386
- [Background] Troster AI, Pahwa R, Fields JA, Tanner CM, Lyons KE. Quality of life in Essential Tremor Questionnaire (QUEST): development and initial validation. Parkinsonism Relat Disord. 2005 Sep;11(6):367-73. doi: 10.1016/j.parkreldis.2005.05.009. PMID 16103000
- See also: Prescribing information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2015/206406s001lbl.pdf